CLINICAL TRIAL: NCT00903461
Title: Safety and Efficacy Evaluation of Radiation and Cetuximab Plus Intratumoral EGFR Antisense DNA Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Safety and Efficacy of Radiation/Cetuximab Plus EGFR Antisense DNA for Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: drug supply issues
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-121; 1R21CA130241-01A1 (NIH)
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck; Squamous Cell Carcinoma of the Head and Neck; Squamous Cell Carcinoma, Head And Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EGFR Antisense DNA (Experimental): EGFR AS will be administered by direct intratumoral injection using direct visualization, endoscopy, or imaging-guidance (ultrasound) as clinically determined. Subjects will receive a total of up to 7 weekly intratumoral injections of EGFR antisense (or less if there is no identifiable tumor) starting 2 weeks prior to radiation. Patients will receive a total EGFR AS dose of 1.92 milligrams in 1.78 milliliters on each weekly treatment. This dose may be delivered equally in the same tumor site per weekly session, the primary tumor or cervical lymph nodes.
  Interventions: Biological: EGFR Antisense DNA

INTERVENTIONS:
Biological: EGFR Antisense DNA — * Intratumoral EGFR AS injections weekly x 7 weeks (or less if there is no identifiable tumor), starting 2 weeks prior to radiation. The first EGFR AS injection must be given after cetuximab is administered. Subsequent EGFR AS injections can be given before or after cetuximab is administered. Injections will be in the primary and/or lymph nodes. One site will be injected per weekly session. If it is necessary the antisense injection can be scheduled within 1 business day of the original schedule date and then resume the original schedule
  * EGFR AS will be administered by direct intratumoral injection using direct visualization, endoscopy, or imaging-guidance (ultrasound) as clinically determined. The same lesion (primary tumor or lymph node) will be injected during treatment.

SUMMARY:
The Epidermal Growth Factor Receptor (EGFR) is highly expressed in SCCHN and its overexpression is associated with poor patient outcome. EGFR is a promising target of anticancer therapy. We have developed EGFR antisense DNA as a safe and potentially efficacious treatment for SCCHN as shown in a previous phase I study conducted at the University of Pittsburgh. Cetuximab (Erbitux or C225) is a chimerized EGFR monoclonal antibody that has produced positive results in a phase III trial in SCCHN when added to radiation therapy and was approved by the FDA for the treatment of locally advanced SCCHN. Radiation plus cetuximab is considered a standard treatment, especially for patients who are not good candidates for chemotherapy. In the current study, we plan to evaluate the addition of intratumoral EGFR antisense DNA (EGFR AS) to standard radiation with concurrent cetuximab in patients.

DETAILED DESCRIPTION:
Subject population We will enroll patients with SCCHN who are suitable for intratumoral injections of EGFR antisense. Please see eligibility criteria.

Treatment plan

EGFR AS will be administered by direct intratumoral injection using direct visualization, endoscopy, or imaging-guidance (ultrasound) as clinically determined . Patients will receive a total of up to 7 weekly intratumoral injections of EGFR antisense (or less if there is no identifiable tumor) starting 2 weeks prior to radiation. Patients will receive standard radiation 70 Gy/200 cGy/daily, 5 days/week,excluding weekends and holidays, with concurrent cetuximab 250 mg/m2, after a loading dose of 400 mg/m2 2 weeks prior to starting radiation.

Statistical Design and Sample Size The study will be conducted in two-stages. In the first stage, 11 patients with stage IVA-C or recurrent disease will be evaluated for safety. If the regimen is deemed safe, a total of 31 patients with stage III or IVA-B, previously untreated SCCHN will be enrolled in the second stage of the study.

ELIGIBILITY:
3.1 Eligibility Criteria

* First stage Patients with current AJCC edition stage IVA-IVC or recurrent or metastatic head and neck cancer will be eligible. Patients with M1 disease must have asymptomatic or low volume distant metastasis and require palliation for local and regional disease
* Second stage (phase II part) Patients with current AJCC edition stage III-IVB (T1-T4, N1-3M0) head and neck cancer, except WHO type II and III nasopharyngeal cancer, including unknown primary tumors.
* Histologically or cytologically confirmed diagnosis of squamous cell carcinoma or variants or poorly differentiated carcinoma.
* Unidimensionally measurable disease (RECIST criteria).
* ECOG Performance Status of 0-2
* In the second stage of the study, therapy will be administered with a curative intent and patients should not have recurrent disease or distant metastasis.
* Primary tumor and/or lymphadenopathy should be technically suitable for intratumoral injections. The Otolaryngologist specialist on the head and neck team will determine this feasibility.
* Participating patients should agree to undergo a tumor biopsy at baseline as well as approximately 2 weeks later as specified in study schema.
* Prior treatment

  * First stage: any prior treatment, except prior therapy which specifically and directly targets the EGFR pathway, administered within the last 6 months. No prior radiation therapy to the head and neck.
  * Second stage: no prior chemotherapy, biologic/molecular targeted therapy (including any prior therapy which specifically and directly targets the EGFR pathway), or radiotherapy for head and neck cancer.
* Prior surgical therapy will consist only of incisional or excisional biopsy, including tonsillectomy, and organ sparing procedures, including neck dissection. Any non-biopsy surgical procedure for head and neck cancer must have taken place at least one month before initiating protocol treatment, at the treating physician's discretion.
* Patients must have organ and marrow function as defined below:

Absolute neutrophil count >/=1,000/µL

Platelets >/=75,000/µL

Hemoglobin >/= 10 g/dL

Total bilirubin <2 x upper normal institutional limits

Creatinine clearance > 20 mL/min

* Age of >/= 18 years
* Because radiation therapy is known to be teratogenic and EFGR inhibitors may have teratogenic potential, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation, and for 3 months after completing study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document.

3.2 Exclusion Criteria

* Severe renal insufficiency (creatinine clearance < 20 mL/min)
* Treatment with anticoagulants, except when used to maintain the patency of a central venous line, or INR >1.5, or PTT ratio >1.5.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements. Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure.
* Patients may not be receiving any other investigational agents.
* No history of prior malignancy, with the exception of curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer, DCIS or LCIS of the breast, localized early stage prostate cancer, or malignancy that has been treated with a curative intent with a 3-year disease-free survival.
* Pregnant women are excluded from this study because cetuximab, EGFR AS, and radiation have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cetuximab and EGFR AS, breastfeeding should be discontinued if the mother is treated with cetuximab. The effects of cetuximab and EGFR AS on the developing human fetus at the recommended therapeutic dose are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while in this study, she should inform her treating physician immediately.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible drug interactions with cetuximab. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated. . HIV status of the patient will be obtained from the patient's history via discussion with the investigator. HIV testing is not required.
* Prior severe infusion reaction to a monoclonal antibody.
* Patients who are not informed of and are not willing to comply with the investigational nature of the study and have not signed a written informed consent in accordance with institutional and good clinical practice guidelines.
* Phase 2 ONLY (second stage) - Subjects with M1 disease will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Disease progression | baseline, 4, 7, 10, and 13 months after study treatment.
  Change in tumor size based on CT or MRI scans of the same tumor(s) of the head and/or neck as compared to baseline measurement.

SECONDARY OUTCOMES:
Number of adverse events associated with study treatment | 2 weeks
Response rate | baseline, 4, 7, 10, and 13 months after study treatment.
  Change in tumor size based on CT or MRI scans of the same tumor(s) of the head and/or neck as compared to baseline measurement.
Determine the effect of EGFR antisense therapy on EGFR and EGFR-related biomarkers. | 3 years
Examine the transfection of the EGFR antisense gene therapy in vivo. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bauman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States